CLINICAL TRIAL: NCT03743779
Title: Mastering Diabetes Pilot Study
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Other Study IDs: 18-X-272
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; lifestyle; plant-based, whole food; vegetarian; vegan; exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Participants enrolled in Mastering Diabetes.
  Interventions: Behavioral: Mastering Diabetes

INTERVENTIONS:
Behavioral: Mastering Diabetes — The Mastering Diabetes provides a step-by-step program to transition to a low-fat, plant-based, whole-food lifestyle and reduce overwhelm. The program also provides direct access to expert coaches in the online community, which contains others living with all forms of diabetes. I includes access to live Q&A videoconferences twice per month to interact with coaches and personalize the experience.
  The program is designed with seven core modules. Many participants continue in the program after completion of the modules for ongoing support.
  The cost was $29/month or $249/year, but as of July 2018, only the $249/year option is offered.

SUMMARY:
This is a pilot study looking at past results of the Mastering Diabetes program utilizing a survey.

DETAILED DESCRIPTION:
Adult past and present participants of Mastering Diabetes will be sent an email asking for their participation in the survey. The email will contain a hot link to a REDCap survey which will begin with a description of the study followed by a consent form. Once the consent is agreed, the survey will ask for participants' demographics and information about the variables described below

No personal identifiable information is being collected.

The data from this study will help develop a prospective study to better evaluate the effectiveness of Mastering Diabetes in controlling diabetes.

Future comparative studies between programs are anticipated, which will help identify the strengths and weaknesses of different programs, as well as identify subpopulations that might benefit from one program as opposed to another.

Data will be shared via posters and papers among the lifestyle medicine community to help contribute to better lifestyle interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adult past and present participants of Mastering Diabetes

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with diabetes who enroll in the Mastering Diabetes program
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin | 1 year
  change in glycosylated hemoglobin during program
weight | 1 year
  change in weight during the program

SECONDARY OUTCOMES:
perception of health change | 1 year
  Survey question is:
  Since completing Mastering Diabetes:
  1. My health has continued to improve
  2. My health has neither improved or declined
  3. My health has declined
  4. I don't know if my health has improved or declined
perception of benefit | 1 year
  Survey question is:
  I feel that Mastering Diabetes was:
  1. Very helpful
  2. Somewhat helpful
  3. Neither helpful or unhelpful
  4. Somewhat unhelpful
  5. Very unhelpful
adherence | 1 year
  Survey question:
  Concerning the changes I made during participation in Mastering Diabetes:
  1. I am still doing all of them
  2. I am still doing most of them
  3. I am still doing about half of them
  4. I am still doing some of them
  5. I am not doing any of them

CONTACTS AND LOCATIONS:
Overall Officials: David Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided